CLINICAL TRIAL: NCT00418483
Title: A Sequential Phase I/II Dose Escalation and Dose Selection Safety Study of Regional Intra-thrombus Plasmin (Human) Infusion In Acute Lower Extremity Native Artery or Bypass Graft Occlusion
Brief Title: A Dose Escalation and Safety Study of Plasmin (Human) In Acute Lower Extremity Native Artery or Bypass Graft Occlusion
Acronym: PRIORITY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050003
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Arterial Occlusive Diseases
Keywords: thrombolytic; thrombolysis; acute peripheral arterial occlusion; peripheral vascular disease; thrombosis; endovascular
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Vascular Diseases; Thrombosis | interventions — Fibrinolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Plasmin (Human) 25 mg (Experimental): Plasmin (Human) 25 mg
  Interventions: Biological: Plasmin (Human) 25 mg
- Plasmin (Human) 50 mg (Experimental): Plasmin (Human ) 50 mg
  Interventions: Biological: Plasmin (Human) 50 mg
- Plasmin (Human) 75 mg (Experimental): Plasmin (Human) 75 mg
  Interventions: Biological: Plasmin (Human) 75 mg
- Plasmin (Human) 100 mg (Experimental): Plasmin (Human) 100 mg
  Interventions: Biological: Plasmin (Human) 100 mg
- Plasmin (Human) 125 mg (Experimental): Plasmin (Human) 125 mg
  Interventions: Biological: Plasmin (Human) 125 mg
- Plasmin (Human) 150 mg (Experimental): Plasmin (Human) 150 mg
  Interventions: Biological: Plasmin (Human) 150 mg
- Plasmin (Human) 175 mg (Experimental): Plasmin (Human) 175 mg
  Interventions: Biological: Plasmin (Human) 175 mg

INTERVENTIONS:
Biological: Plasmin (Human) 25 mg — Plasmin (Human) 25 mg delivered via an infusion catheter into the thrombus over approximately 5 hours.
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: Plasmin (Human) 25 mg
Biological: Plasmin (Human) 50 mg — Plasmin (Human) 50 mg delivered via an infusion catheter into the thrombus over approximately 5 hours.
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: Plasmin (Human) 50 mg
Biological: Plasmin (Human) 75 mg — Plasmin (Human) 75 mg delivered via an infusion catheter into the thrombus over approximately 5 hours.
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: Plasmin (Human) 75 mg
Biological: Plasmin (Human) 100 mg — Plasmin (Human) 100 mg
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: Plasmin (Human) 100 mg
Biological: Plasmin (Human) 125 mg — Plasmin (Human) 125 mg delivered via an infusion catheter into the thrombus over approximately 5 hours.
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: Plasmin (Human) 125 mg
Biological: Plasmin (Human) 150 mg — Plasmin (Human) 150 mg delivered via an infusion catheter into the thrombus over approximately 5 hours.
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: Plasmin (Human) 150 mg
Biological: Plasmin (Human) 175 mg — Plasmin (Human) 175 mg delivered via an infusion catheter into the thrombus over approximately 5 hours.
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: Plasmin (Human) 175 mg

SUMMARY:
The purpose of this study is to evaluate the safety of increasing doses of intra-thrombus Plasmin (Human) in acute peripheral arterial occlusion (aPAO). The ability of these Plasmin doses to dissolve the clots will be estimated by arteriography.

DETAILED DESCRIPTION:
There is an unmet need for proven thrombolytic agent in acute peripheral arterial occlusion (aPAO). The current assortment of plasminogen activators are slow to dissolve clots in the leg, and may lead to bleeding complications. Plasmin is a direct thrombolytic that may act more quickly when infused directly into the clot and thus assist in restoring blood flow to the leg. There is a large reserve in blood alpha-2 antiplasmin in the blood to rapidly inactivate Plasmin outside of the clot. Plasmin has the potential for an improved bleeding risk profile in aPAO.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Women of childbearing potential must use adequate contraception for the duration of the study and must have a negative pregnancy test prior to study entry.
* Unilateral limb ischemia: SVS acute ischemia Category I or IIa.
* Onset of symptoms </= 14 days.
* Thrombosed (non-embolic) infrainguinal graft (synthetic, autologous, or single outflow composite) or infrainguinal native artery. For native arteries, only occlusions of ≥ 10 cm in length are eligible.
* Diagnosis of occlusive thrombus in the graft or artery by arteriography after Informed Consent is obtained.
* Ability to traverse the thrombus with a guidewire.
* Signed informed consent prior to study entry.

Exclusion Criteria:

* Clinical evidence of significant disease that may interfere with the patient successfully completing the trial.
* Women who are pregnant or lactating, or first 10 days post-partum.
* Previous hemorrhagic stroke at any time. Thrombotic or embolic stroke or cerebrovascular events (including transient ischemic attack (TIA)) within one year.
* Intracranial or spinal neuro-surgery, or severe intracranial trauma in the last 3 months. Major surgery, organ biopsy, or major trauma within the last 10 days. Lumbar puncture or non-compressible arterial puncture in the last 10 days. Intra-ocular surgery within the last 10 days.
* Current bleeding diathesis. Active gastrointestinal or organ bleeding. Minor bleeding such as normal menses, cystitis, or minor hemorrhoidal bleeding are not exclusions.
* Uncontrolled arterial hypertension, defined as a systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg.
* Known intracranial neoplasm, aneurysm, or arterio-venous malformation.
* Platelet count < 75 x 10e9/L.
* Occlusion of a graft within 6 months of placement.
* Medically unable to tolerate an open vascular procedure.
* Known prothrombotic condition.
* Hemoglobin <10.0 g/dL
* Impaired renal function or renal disease that constitutes a contraindication to contrast angiography, including creatinine > 2.0 mg/dL or subjects on renal dialysis.
* Treatment with a glycoprotein IIb/IIIa class of platelet inhibitor within the past 5 days, for example, abciximab (ReoPro®), eptifibatide (Integrilin®) or tirofiban (Aggrastat®).
* Treatment with warfarin (Coumadin®) and with an INR of >1.7 (elevated INR at screening may be corrected prior to study enrollment.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Thrombolysis | Approximately 5 hours after start of treatment
  Thrombolysis at the end of treatment compared to baseline by arteriography

SECONDARY OUTCOMES:
Thrombolysis | Approximately 2 hours after start of treatment
  Thrombolysis at 120 minutes compared to baseline by arteriography
Avoidance of open surgical procedures | 30 days
  Percent of subjects at Day 30 who avoid open surgical procedures
Avoidance of amputation | 30 days
  Percent of subjects at Day 30 who avoid amputation
Avoidance of additional catheter-directed thrombolysis with a plasminogen activator or mechanical device thrombectomy | 30 days
  Percent of subjects at Day 30 who avoided additional catheter-directed thrombolysis with a plasminogen activator or mechanical device thrombectomy.
Avoidance of both open surgical procedures and additional thrombolysis with a plasminogen activator or mechanical device thrombectomy. | 30 days
  Percent of subjects at Day 30 who avoided both open surgical procedures and additional thrombolysis with a plasminogen activator or mechanical device thrombectomy.
Physiologic reperfusion defined as improvement in ankle brachial index (ABI) | End of treatment, post intervention procedures, Day 1 to 2, Day 7, and Day 30
  Physiologic reperfusion defined as improvement in ABI (increase of ≥ 0.15) determined at the end of treatment, post intervention procedures, Day 1 to 2, Day 7, and Day 30.
Patency assessed by duplex ultrasound imaging | Day 7 and Day 30
  Patency assessed by duplex ultrasound imaging on the affected leg on Day 7 and Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Comerota, MD, Principal Investigator — Jobst Vascular Center
Locations (1):
- Jobst Vascular Institute, Toledo, Ohio, United States